CLINICAL TRIAL: NCT03941821
Title: The Efficacy, Safety and Long-term Prognosis of Glecaprevir/Pibrentasvir in the Treatment of Chronic Hepatitis C Patients in China--A Real-world Study
Brief Title: Glecaprevir/Pibrentasvir Real-world Study in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: G/P RWS China
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Chronic Hepatitis c
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, urine and whole blood will be restored in central lab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- G/P treatment: Chronic hepatitis C patients who will recieve Glecaprevir/Pibrentasvir treatment
  Interventions: Drug: Glecaprevir/Pibrentasvir

INTERVENTIONS:
Drug: Glecaprevir/Pibrentasvir — Chronic hepatitis C patients will be given Glecaprevir/Pibrentasvir treatment
  Other Names: Mavyret

SUMMARY:
To evaluate the efficacy, adverse effect, short - and long-term outcomes of Glecaprevir/Pibrentasvir for the treatment of chronic hepatitis C (non-cirrhotic or compensatory cirrhosis)in China through a real-world study

DETAILED DESCRIPTION:
This study is a multi-center, prospective, real-world study, aiming to investigate the use of Glecaprevir/Pibrentasvir in routine clinical management of chronic hepatitis C patients and evaluate its effectiveness and safety across a heterogeneous population in China.Approximately 800 patients will take part in this study, 20 sites will be included which distribute in China's major cities, thus each site will enroll 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Meet the standard of Glecaprevir/Pibrentasvir treatment

Exclusion Criteria:

* Patients have contraindications to Glecaprevir/Pibrentasvir
* Pregnancy or lactation
* Malignancy
* Decompensatory cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C who will received Glecaprevir/Pibrentasvir treatment and meet the inclusion and exclusion criteria above
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-06-30 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
SVR 12 | 12 weeks after Glecaprevir/Pibrentasvir treatments
  The effectiveness of Glecaprevir/Pibrentasvir treatments and SVR rate 12 weeks after Glecaprevir/Pibrentasvir treatments
progression of Chronic liver disease | 5 years after Glecaprevir/Pibrentasvir treatments
  Incidence of liver disease progression (such as cirrhosis, decompensation of liver function, liver cancer, liver transplantation, or liver related death)

SECONDARY OUTCOMES:
long term outcome | 5 years
  Assess the duration of the virologic response (5 years) in CHC patients with daas-based regimens who have achieved a sustained virologic response (svr12/24) at 12 or 24 weeks after the end of treatment and analyze the factors influencing the recurrence of HCV
HRQOL | 5 years
  To evaluate the impact of DAAs treatment on health-related quality of life (HRQOL) and health status of CHC patients

CONTACTS AND LOCATIONS:
Overall Officials: Qin Ning, PHD,MD, Study Chair — Department and Institute of Infectious Disease, Tongji Hospital, Tongji Medical College HUST